CLINICAL TRIAL: NCT02102048
Title: ATAGLU: Study of Glucose Metabolism in HIV Positive Patients That Switch From Another Protease Inhibitor to Boosted or Unboosted Atazanavir
Brief Title: ATAGLU: Study of Glucose Metabolism in HIV Positive Patients That Switch From Another Protease Inhibitor to Atazanavir
Acronym: ATAGLU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giancarlo Ceccarelli, MD, PhD, MSc, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPHID-UniRoma02
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: HIV
Keywords: HIV; diabetes; glucose metabolism; antiretroviral therapy; ritonavir; atazanavir
MeSH Terms: conditions — Diabetes Mellitus | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atazanavir (Active Comparator): patients that switch cART to boosted or unboosted ATV
  Interventions: Drug: Atazanavir
- other Protease Inibithors (No Intervention): patients that continue the previous cART without changes.

INTERVENTIONS:
Drug: Atazanavir
  Other Names: Reyataz
  Arms: Atazanavir

SUMMARY:
The association between HIV infection , insulin resistance and diabetes mellitus is the topic of many studies that have attempted to analyze the problem from different points of view. In fact, the risk of insulin resistance in HIV-positive patients on antiretroviral therapy seems to depend not only on the same factors that determine its incidence in the general population , but also on the effects of antiretroviral therapy on glucose metabolism. To confirm this observation, studies that have evaluated the incidence of diabetes in patients with HIV infection on antiretroviral therapy have shown that the incidence of diabetes in infected individuals is significantly higher than that observed in the uninfected population. Moreover others preliminar stadies observed that protease inhibitors may induce hyperglycemia and diabetes mellitus. Anyway at this moment no large data are available that indicate the utility to modify the antiretroviral therapy in HIV positive patients with a damage of glucose metabolism.

ATAGLU is a cohort composed by HIV positive patients in effective and stable combined antiretroviral therapy (cART) with undetectable viral load. All patients studied had carried out a therapy with Lopinavir/Ritonavir (LPV/r) + optimal backbone therapy (OBT) and then in part switch to Atazanavir (ATV) + OBT or Atazanavir/ritonavir (ATV/r) + OBT , in part continue with LPV/r + OBT .

The objective was to characterize the changes of carbohydrate profile of a cohort of patients who made a switch from a regimen with LPV/r to boosted or unboosted ATV.

ELIGIBILITY:
Inclusion Criteria:

* HIV postive patients
* Patients on stable and effective antiretroviral therapy with a Protease Inhibitor

Exclusion Criteria:

* use of Atazanavir before the enrolment
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Homeostatis Model Assessment-Insulin Resistance (HOMA-IR) value | 1 year
  difference between Homeostatis Model Assessment-Insulin Resistance (HOMA-IR) value of patients that continue cART with LPV/r and patients that switch to ATV/r or ATV

SECONDARY OUTCOMES:
insulinemia | 1 year
  difference between insulinemia value of patients that continue cART with LPV/r and patients that switch to ATV/r or ATV

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Vullo, MD, Principal Investigator — University of Rome "Sapienza" (Italy)
Locations (1):
- Department of Public Heath and Infectious Diseases. University of Rome "Sapienza" (Italy), Rome, Italy